CLINICAL TRIAL: NCT03789747
Title: Incidence and Risk Factors of Acute Kidney Injury After Craniotomy: a Single-Center Experience
Brief Title: Acute Kidney Injury After Craniotomy
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Jianfang Zhou, Principal investigator, Beijing Tiantan Hospital
Other Study IDs: Beijing Tiantan Hospital
Record Dates: First submitted 2017-05-11; First posted 2018-12-31 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-02

CONDITIONS: Epidemiology; Acute Kidney Injury; Risk Factor
Keywords: incidence; prognosis; acute kidney injury; risk factor; post-craniotomy
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: As a observational study, there is no intervention. — As a observational study, there is no intervention.

SUMMARY:
The aim of this study was to investigate the incidence, risk factors and prognosis of acute kidney injury (AKI) in critically ill patients after craniotomy.

DETAILED DESCRIPTION:
This was a prospective, single-center, cohort study that included adult patients who were admitted to the ICU of Beijing Tiantan Hospital from January 2017 to December 2018 after craniotomy and had a stay in the ICU for ≥ 24 hours (patients with preoperative AKI were excluded). Data collected included patient demographics (age, gender, underlying diseases, baseline serum creatinine, etc.), primary diagnosis, perioperative information, disease severity scores, as well as the occurrence of hypernatremia and hyperchloremia within 48 hours after ICU admission. For patients with AKI, pre-AKI sepsis and shock, and the recovery of renal function were recorded. All patients were followed until discharge, and information about prognosis was recorded. Multivariate regression analysis was used to identify the risk factors of AKI.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent craniotomy
* admitted into ICU ward and the ICU length of stay ≥24h

Exclusion Criteria:

* Age< 18 years;
* Patients with pre-existing acute kidney injury (AKI) and chronic kidney disease undergoing long-term renal replacement therapy (RRT) .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent craniocerebral operation and admitted into intensive care unit (ICU) between January 2017 and December 2018 were consecutively screened. Patients developed AKI after ICU admission were deemed as cases, and those without AKI were included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence and outcome of AKI after Craniotomy | during hospitalization
  All adult patients who underwent craniotomy and admitted into intensive care unit (ICU) between January 2017 and December 2018 were screened for acute kidney injury.

SECONDARY OUTCOMES:
Risk factors for AKI after Craniotomy | during hospitalization
  Logistic regression analysis was employed to assess the risk factors for AKI. Variables with a significance level of P<0.2 in univariate analysis and clinical relevance were included as adjustment factors in the regression analysis model. The calibration of the model was evaluated using the Hosmer-Lemeshow goodness-of-fit test.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxin Zhou, MD, Study Director — Beijing Tian Tan Hospital; Guangzhi Shi, MD, Study Director — Beijing Tian Tan Hospital
Locations (1):
- Beijing Tian Tan hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No